## Use of Repetitive Transcranial Magnetic Stimulation to Augment Hypnotic Analgesia

Statistical Analysis Plan

NCT02969707

January 4, 2024

Data were collected and organized using the REDCap methodology, and analysis was performed in the SPSS v.26.0 environment. According to our preregistered plan, analyses were completed within the intention-to-treat principle, and reported P values are nominal. To test the change in HIP scores following SHIFT, pre- to post-SHIFT changes in HIP scores ( $\Delta$ HIP) were calculated by subtracting the immediate post-spaced SHIFT score from the pre-spaced SHIFT score. Neither the pre- or post-spaced SHIFT HIP variables nor the  $\Delta$ HIP scores met the criteria for the assumption of normality (all Shapiro—Wilk P values < 0.001), rendering the first step in our preregistered plan of testing our hypotheses using analysis of variance (ANOVA) inappropriate. As such, we used non-parametric tests; within-group pre/post-SHIFT changes in HIP scores were tested using a two-tailed Wilcoxon signed-rank test. Two-tailed Mann—Whitney U-tests were used for group comparisons of  $\Delta$ HIP scores between the active and sham groups. Effect sizes for the non-parametric tests were calculated using Cohen's r statistic. The study blind was tested using the chi-squared test.